CLINICAL TRIAL: NCT06088433
Title: Safety and Efficacy of Ticagrelor Single Antiplatelet Therapy in Patients With High Risk of Bleeding After Drug-coated Balloons for Coronary Small Vessel Disease: A Prospective, Randomized, Open-label, Blinded-endpoint Evaluation, Single-center Study
Brief Title: Ticagrelor Single Antiplatelet Therapy in Patients With High Risk of Bleeding After DCB for Coronary Small Vessel Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Qian Haiyan, MD, PhD, Fu Wai Hospital, Beijing, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-I2M-C&T-B-050
Record Dates: First submitted 2023-06-07; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Coronary Heart Disease
Keywords: CHD; DCB; SAPT; Ticagrelor
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPT (Experimental): Ticagrelor SAPT 90mgBID for 1 month, followed by 60mgBID
  Interventions: Drug: Ticagrelor
- DAPT (Active Comparator): Aspirin 100mgQD+Clopidogrel 75mgQD for 1 month, followed by clopidogrel 75mgQD
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — Comparison of 12 month of ticagrelor SAPT（90mgBID*1 month, followed by 60mgBID) versus 12 months of dual anti-platelet therapy (Aspirin 100mgQD+clopidogrel 75mgQD * 1 month, followed by clopidogrel 75mgQD)
  Other Names: Brilinta/Brilique
  Arms: SAPT
Drug: Clopidogrel — Comparison of 12 month of ticagrelor SAPT（90mgBID*1 month, followed by 60mgBID) versus 12 months of dual anti-platelet therapy (Aspirin 100mgQD+clopidogrel 75mgQD * 1 month, followed by clopidogrel 75mgQD)
  Arms: DAPT
Drug: Aspirin — Comparison of 12 month of ticagrelor SAPT（90mgBID*1 month, followed by 60mgBID) versus 12 months of dual anti-platelet therapy (Aspirin 100mgQD+clopidogrel 75mgQD * 1 month, followed by clopidogrel 75mgQD)
  Other Names: Acetylsalicylic Acid
  Arms: DAPT

SUMMARY:
The present study is aimed to determine the safety and efficacy of Ticagrelor single antiplatelet therapy (SAPT) in patients with primary coronary small vessel disease at high risk of bleeding after drug coated balloon (DCB) therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, blinded-endpoint evaluation, single-center Study. There will be 234 patients with high-risk bleeding and primary coronary small vessel disease after DCB enrolled in our research, randomly dividing into an experimental group (Ticagrelor SAPT, 90mg BID * 1 month, followed by 60mg BID, n=117) and a control group (DAPT, aspirin 100mg QD+clopidogrel 75mg QD * 1 month, followed by clopidogrel 75mg QD, n=117).The primary endpoint is 12 months of Major adverse cardiovascular events (MACE), including death, myocardial infarction, stroke, and target vessel revascularization. The key secondary endpoint is MACE at 1 month. The safety endpoint is BARC bleeding at all levels. Follow up will be conducted at 1 month and 12 months, and platelet inhibition rate will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. CHD patients aged 18-80 with clear indications for PCI, regardless of gender;
2. Received DCB treatment with only one small coronary artery (diameter 2.0-2.75mm);
3. High risk of bleeding (ARC high risk criteria for bleeding): Meets at least one main criterion (use of anticoagulants, liver dysfunction, tumors, history of gastrointestinal bleeding, history of peptic ulcers, creatinine clearance rate<30mL/min, hemoglobin<11g/L, platelet count<100 × 109/L) or 2 sub criteria (age ≥ 75 years old, creatinine clearance rate<60mL/min, history of stroke/TIA, hemoglobin 11-12.9g/L for males or 11-11.9g/L for females);
4. Willing to participate in trials and complete follow-up;
5. Signed an informed consent form approved by the Ethics Committee;

Exclusion Criteria:

1. Simultaneously or plan to perform other coronary PCI procedures in batches, including stent implantation, DCB treatment for non-small vessel lesions, and DCB treatment for in stent restenosis lesions.
2. High ischemic risk: a. ACS within 1 year; b. Perform stent implantation or CABG surgery within 1 year; c. Double or multi vessel lesions rearched incomplete revascularization; d. In addition to the target lesions for DCB intervention, there are other stenosis ≥ 90%, regardless of whether PCI is planned or not;
3. Anticoagulant drugs are required for atrial fibrillation/deep vein thrombosis (including pulmonary embolism)/mechanical valve implantation;
4. Cardiomyopathy (HCM/DCM/RCM);
5. Severe ventricular arrhythmias requires radiofrequency ablation or ICD implantation;
6. Chronic obstructive pulmonary disease (bronchial asthma, chronic bronchitis, emphysema, pulmonary heart disease);
7. Serious infectious diseases, including active hepatitis B, hepatitis C or AIDS patients;
8. Blood system diseases with coagulation disorders such as thrombocytopenia, leukemia, and hemophilia;
9. Thrombotic diseases such as antiphospholipid antibody syndrome;
10. Cognitive impairment;
11. Not willing to participate in experiments or cooperate with follow-up;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 12 months after randomization
  A composite of mortality, non-fatal myocardial infarction, non-fatal stroke or target vessel revascularization

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (Key secondary endpoint) | 1 month after randomization
  A composite of mortality, non-fatal myocardial infarction, non-fatal stroke or target vessel revascularization
Platelet inhibition rate (thromboelastogram) | 12 months after randomization
Rate of patients taking medicine as prescribed | 12 months after randomization
Rate of patients discontinued medication due to bleeding | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Qian, MD, PhD, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China